CLINICAL TRIAL: NCT02540421
Title: Presence of Positive Resection Margins, Hypooestrogenism and Specimen Volume May Influence Risk of Disease Recurrence in Patients With High-grade Cervical Intra-epithelial Neoplasia Undergoing Large Loop Excision of the Transformation Zone
Brief Title: Recurrence in High-grade Lesions After Conization
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Emerson Oliveira, PhD, Faculdade de Medicina do ABC
Other Study IDs: CIN1701
Record Dates: First submitted 2014-10-15; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: cervical intraepithelial neoplasia; human papillomavirus; conization
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Recurrent lesions
- Control: Absence of lesions

SUMMARY:
Objectives: To identify factors associated with disease recurrence in patients with high-grade cervical intra-epithelial neoplasia (CIN) undergoing large loop excision of the transformation zone (LLETZ).

Study Design: A case-control study that included 103 patients. Patients were included in the study if they had a history of surgery for conization by LLETZ for the histopathological diagnosis of cervical intraepithelial neoplasia grades II and III (CIN II and CIN III). Follow-up exams were conducted every six months with Pap smear collection and colposcopic examination with biopsy, when necessary, for a minimum period of twelve months. Cure was defined as a normal follow-up examination within 24 months. During follow-up, relapse occurred when cytology and/or biopsy results showed that CIN had returned after 12 months, at which time a new cervical conization by LLETZ was performed.

ELIGIBILITY:
Inclusion Criteria:

1. history of surgery for conization

Exclusion Criteria:

1. under 18 years of age,
2. immunosuppressed,
3. Patient with a histopathological diagnosis of low-grade intraepithelial neoplasia
4. Patient with invasion, or surgical margins obtained by LLETZ that were unable to be evaluated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were included in the study if they had a history of surgery for conization by LLETZ for the histopathological diagnosis of cervical intraepithelial neoplasia grades II and III (CIN II and CIN III).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2001-01; Primary Completion 2007-01 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Recurrence rates after conization | 12 months
  Number of patients who are regarded as recurrence based on the following criteria:
  - relapse occurred when cytology and/or biopsy showed that CIN had returned after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: EMERSON OLIVEIRA, PhD, Principal Investigator — FACULTY OF MEDICINE OF ABC
Locations (1):
- Emerson de Oliveira, Santo André, São Paulo, Brazil